CLINICAL TRIAL: NCT00002313
Title: Extended Maintenance Protocol for Phase I/II Clinical Study of Nystatin I.V. (Intravenous) in Patients With HIV Infection (NOTE: Continuation Study Intended Only for Patients Who Have Completed FDA 103B)
Brief Title: A Study of Nystatin in HIV-Infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Argus Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 103C; AR-91-35,606-005A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1994-04

CONDITIONS: HIV Infections
Keywords: Nystatin; Didanosine; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Nystatin; Didanosine

INTERVENTIONS:
Drug: Nystatin
Drug: Didanosine

SUMMARY:
To evaluate the clinical toxicity, safety, and potential anti-HIV activity of intravenous nystatin in patients with HIV infection who have completed protocol FDA 103C. To evaluate the safety and potential antiviral activity of intravenous nystatin and oral didanosine (ddI) administered in an alternating regimen in this patient population.

DETAILED DESCRIPTION:
Patients who have completed protocol FDA 103B are offered the option of receiving extended maintenance. Patients who have received no prior ddI are treated either with intravenous nystatin alone (at the same dose level administered in FDA 103B) or with a regimen of intravenous nystatin and ddI alternating on 3-week cycles. Treatment continues for 12 weeks.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Completed 12 weeks of therapy with intravenous nystatin on protocol FDA 103B.
* No evidence of toxicity or progression of disease on protocol FDA 103B. (See protocol FDA 103B for initial entry requirements.)

Active drug or alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Twelve Oaks Hosp, Houston, Texas, United States

REFERENCES:
- [Background] Rios A, Brewton G, Crofoot G, Quesada J, Lenk R, Lopez-Berenstein G. A phase I-II clinical study of Nystatin-LF IV in patients with HIV infections. Int Conf AIDS. 1993 Jun 6-11;9(1):483 (abstract no PO-B26-2089)